CLINICAL TRIAL: NCT00096590
Title: Evaluation of a Novel Blood Test Hypercoagulability in Surgical Patients With Metastatic Carcinoma: A Pilot Study
Brief Title: Detecting Abnormal Blood Clotting in Patients With Metastatic Cancer Undergoing Surgery
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000440092; NCI-05-CC-0033; NCT00464360 (obsolete NCT alias)
Record Dates: First submitted 2004-11-11; First posted 2004-11-12 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2007-06

CONDITIONS: Thromboembolism; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: thromboembolism; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Thromboembolism | interventions — Bleeding Time; Immunoenzyme Techniques

INTERVENTIONS:
Other: coagulation study
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Other: physiologic testing
Procedure: study of high risk factors

SUMMARY:
RATIONALE: A test that detects abnormal blood clotting in patients with cancer may help doctors plan cancer surgery.

PURPOSE: This laboratory study is looking at a new blood test to detect abnormal clotting in patients with metastatic cancer undergoing surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether whole blood thrombin generation assay (WBTGA) detects hypercoagulability in patients with metastatic carcinoma compared with a healthy control group.
* Determine whether results of the WBTGA will change as a result of major surgery performed on patients with metastatic carcinoma.
* Establish a reference interval for the WBTGA using healthy controls.

Secondary

* Compare a battery of plasma components known to affect or reflect coagulant or fibrinolytic reactions in patients with metastatic carcinoma vs healthy controls.
* Establish reference intervals for this battery of tests using healthy controls.
* Determine how major surgery in cancer patients affects this battery of factors.
* Identify changes in these factors that correlate with changes in the WBTGA.
* Compare the results of WBTGA tests in patients who develop venous thromboembolism (VTE) with those who do not.

OUTLINE: This is a pilot study.

Blood samples of patients are collected on day -7 and day 1 after surgery.

Blood samples of healthy controls are collected once.

After collection, blood samples are analyzed for hypercoagulability by whole blood thrombin generation assay. Routine blood tests are performed, as are immunoenzyme techniques for antigenic tissue plasminogen activator and its inhibitor, thrombin-antithrombin complexes, tissue factor, factor VIIa, D-dimer, and glycocalicin.

PROJECTED ACCRUAL: A total of 30 patients and 30 healthy controls will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients meeting the following criteria:

  * Diagnosis of metastatic carcinoma
  * Must be enrolled in 1 of the following surgical protocols:

    * NCI-99-C-0123
    * NCI-00-C-0069
    * NCI-03-C-0085
    * NCI-03-C-0212
* Healthy control participant* meeting the following criteria:

  * No anemia or thrombocytopenia
  * No history of venous thromboembolism (deep vein thrombosis, pulmonary emboli)
  * No history of coronary artery disease or stroke
  * No chronic inflammatory disease
  * No diabetes mellitus
  * Have not smoked tobacco within the past 6 months NOTE: * Selected on the basis of gender and age to match the patients as they are accrued

PATIENT CHARACTERISTICS:

* No symptomatic infections or other acute illness within the past 14 days

PRIOR CONCURRENT THERAPY:

* At least 3 days since prior drugs known to inhibit platelet function
* At least 7 days since prior acetylsalicylic acid
* No concurrent estrogen contraceptives or hormone replacement therapy
* No concurrent anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-11

PRIMARY OUTCOMES:
Incidence of hypercoagulability

SECONDARY OUTCOMES:
Comparison of the results of whole blood thrombin generation assay tests in patients who develop venous thromboembolism with those who do not

CONTACTS AND LOCATIONS:
Overall Officials: McDonald K. Horne, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Result] Horne MK 3rd, Merryman PK, Cullinane AM, Nghiem K, Alexander HR. The impact of major surgery on blood coagulation factors and thrombin generation. Am J Hematol. 2007 Sep;82(9):815-20. doi: 10.1002/ajh.20963. PMID 17570509